CLINICAL TRIAL: NCT04919434
Title: Intervention to Reduce Exposure to Environmental COntaminant (IRECO)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C20-81; 2021-A00215-36 (Registry Identifier: IRECO)
Record Dates: First submitted 2021-05-26; First posted 2021-06-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Exposure
Keywords: intervention study; chemical assessment; personal care product

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Women will be asked NOT to use their own personal care product during the intervention. They will only have to use the substitute one given by the research team
  Interventions: Other: IRECO

INTERVENTIONS:
Other: IRECO — During 5 days, women included in the study will have to only use personal care product distributed by the research team.

SUMMARY:
Main objective The intervention study IRECO aims to (1) modify habits of personal care product use for the participants and (2) evaluate the impact of those modification on urinary concentration for the following compounds: phthalates, phenols and glycol ether.

Secondary objectives:

The secondary objectives of this study aim to evaluate:

1. impact of modification of personal care product on the levels of biomarkers linked to exposure to environmental pollutant other than phthalates phenol and glycol ether (untargeted analysis) and biomarkers related to health (such as inflammatory biomarkers and oxidative stress).
2. hazard perception linked to the exposure to chemical product present in personal care product
3. barriers to change habits allowing to decrease exposure to environmental pollutant on short and long term as well as levers allowing to remove those barriers.

DETAILED DESCRIPTION:
Many chemical compounds are allowed as ingredients in personal care product. Among those substances, phenols, phthalates and some glycol ether are widely detected in personal care product. Few epidemiological studies suggested association between the use of personal care product and higher urinary concentration of parabens, phthalates, bisphenol A and triclosan. In France, studies in general population also show those associations and suggested higher urinary concentration of some glycol ethers in users of cosmetics, (make up, nail polish, nail polish remover), deodorant, and care product (cream, lotion etc.) The intervention study IRECO (Intervention to Reduce Exposure to environmental Contaminant) aims to study the impact of personal care product on exposure levels of compounds from phenol, phthalates and glycol ether. This project will allow to better characterize sources of exposure of those chemical compounds for which deleterious effect on health is suspected. The results of this study will be informative and will allow to bring concrete solutions to the general population who wish to reduce their exposure. The study will also allow to help decision maker in trying to limit exposure to chemical compounds such as phthalates and phenols in daily consumption product. To date, these type of intervention studies were conducted in the USA and no study have been done in France so far where regulation and consumption habits differs from the USA.

The two main objectives of the intervention study IRECO are: (1) modify habits of personal care product use for the participants and (2) evaluate the impact of those modification on urinary concentration for the following compounds: phthalates, phenols and glycol ether.

To meet those objectives, 100 women with the following inclusion criteria will be included in the study : (1) aged between 18 and 30 years, (2) accept to not use personal care product or use only the alternative personal care product distributed by the research team for 5 days, (3) to not have any known allergies to ingredients in the alternative personal care product, (4) to benefit from the French health assurance ; (5) live in the area of Grenoble (France) (6) speak French fluently, (7) have a freezer to store the urine collected.

The study follow-up will include 12 days of measure divided in three phases :

1. - The pre-intervention phase which will last for 3 days and during which the volunteer will (1) collect a sample of each miction with collection tubes given by a field worker, store those urines in her freezer and (2) use an application to collect data on use of personal care product, cleaning product, food drinks and drugs intakes as well as the hour of each miction. At the end of the pre-intervention phase, 24ml of blood will be withdrawn and a semi-structured interview will be conducted aiming to evaluate volunteer's knowledge on the studied compounds, the presence of those compounds in the ingredients of personal care product and the hazard linked to the exposure of those compounds.
2. - The intervention phase will last 5 days during which the volunteers will: (1) stop using her personal care product and use the alternative ones distributed by the research team , (2) collect a sample of each miction with collection tubes given by a field worker, store those urines in her freezer and (3) use an application to collect data on use of personal care product, cleaning product, food drinks and drugs intakes as well as the hour of each miction. At the end of the pre-intervention phase, 24ml of blood will be withdrawn
3. - The post intervention phase will last 4 days during which the volunteers will: (1) collect a sample of each miction with collection tubes given by a field worker, store those urines in her freezer and (2) use an application to collect data on use of personal care product, cleaning product, food drinks and drugs intakes as well as the hour of each miction

2 months after the intervention a fieldworker will go the volunteer's home to conduct a semi-structured interview on her changes in the use of personal care product following her participation into the intervention study IRECO.

ELIGIBILITY:
Inclusion Criteria:

* be a women
* be older than 18 and younger than 30
* accept to not use or use only the substitute personal care product for 5 days
* no know allergy to ingredients in personal care product
* no skin or allergy disease
* have a medical insurance
* live in Grenoble area
* speak french fluently
* have a freezer to store the urine sample for a week

Exclusion Criteria:

* being pregnant
* working in a job manipulating personal care product
* participating in an other study on cosmetics, personal care product, diet or any other study that may affect exposure to the studied chemicals

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2022-06-26 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2027-06-25 (Estimated)

PRIMARY OUTCOMES:
Modification of exposure to phthalates, phenols and glycol ether | follow-up 1 week
  Urinary concentration of phthalates, phenols and glycol ether will be measured in urine sample. Urinary concentration will be measured in the three phases of the study : before intervention (phase 1), during intervention (phase 2) and after intervention (phase 3). The level of urinary concentration will be compared between each phase : phase 1 versus phase 2 and phase 2 versus phase 3.

SECONDARY OUTCOMES:
Modification of exposure other than phthalates, phenols and glycol ether | follow-up 1 week
  An untargeted approach will be conducted where chemical pollutants other than phthalates, phenols and glycol ether will be measured in urines. Urinary concentration of pollutants will be measured in the three phases of the study : before intervention (phase 1), during intervention (phase 2) and after intervention (phase 3). The level of urinary concentration will be compared between : (a) phase 1 and phase 2 and (b) phase 2 and phase 3.
Hazard perception linked to the exposure to chemical product present in personal care product | during the follow-up week.
  A qualitative analysis will be conducted with the data collected during the sociodemographic interview. The analysis will describe the hazard perception of the volunteers linked to the exposure to chemical products present in personal care product.
Barriers to change habits in the use of personal care product | during the follow-up week and 2 months after the intervention
  A qualitative analysis will be conducted with the data collected during the sociodemographic interview. The analysis will describe the barriers to change habits allowing to decrease exposure to environmental pollutant on short and long term as well as levers allowing to remove those barriers.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut pour l'avancée des biosciences IAB (U1209)/hôpital couple enfant du CHU Grenoble-Alpes, Grenoble, France